CLINICAL TRIAL: NCT07276919
Title: Perioperative Tamsulosin for Treating Voiding Dysfunction Following Prostate Biopsy: A Multicenter, Randomized, Controlled, Open-Label Study
Brief Title: Perioperative Tamsulosin for Treating Voiding Dysfunction Following Prostate Biopsy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University First Hospital Miyun Hospital (Unknown); Taiyuan Central Hospital of Shanxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20251018
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Acute Urinary Retention; LUTS(Lower Urinary Tract Symptoms)
Keywords: acute urinary retention; LUTS(Lower urinary tract symptoms); tamsulosin; prostate biopsy
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin Group (Experimental): The experimental group will receive Tamsulosin Hydrochloride Sustained-Release Capsules (0.2 mg, once daily at night) starting 3 days before the biopsy and continuing until the 6th day after the procedure (10 doses total).
  Interventions: Drug: Tamsulosin 0.2mg
- Control Group (No Intervention): Participants will not receive Tamsulosin during the perioperative period but will undergo the standard prostate biopsy procedure.

INTERVENTIONS:
Drug: Tamsulosin 0.2mg — The experimental group will receive Tamsulosin Hydrochloride Sustained-Release Capsules (0.2 mg, once daily at night) starting 3 days before the biopsy and continuing until the 6th day after the procedure (10 doses total).
  Other Names: Tamsulosin Hydrochloride Sustained-Release Capsules
  Arms: Tamsulosin Group

SUMMARY:
The goal of this clinical trial is to learn if the drug Tamsulosin Hydrochloride works to treat urination difficulties after a prostate biopsy in men.The main questions it aims to answer are:

* Does Tamsulosin Hydrochloride lower the rate of Acute Urinary Retention (inability to urinate) after a prostate biopsy?
* Does Tamsulosin Hydrochloride improve participants' urination symptoms, quality of life, urine flow rate, and post-void residual urine volume?

Researchers will compare the drug group to a control group (receiving no preventive medication) to see if Tamsulosin Hydrochloride works to prevent urination problems.

Participants will:

* Be randomly assigned to either take Tamsulosin Hydrochloride or receive no preventive medication.
* If in the drug group, take one capsule of Tamsulosin Hydrochloride every night, starting 3 days before the biopsy and continuing until 6 days after the biopsy (10 doses total).
* Undergo a standard prostate biopsy procedure (either through the rectum or perineum).
* Return to the clinic 7 days after the biopsy for a follow-up checkup, which will include questions about their symptoms (IPSS and QoL scores) and tests to measure urine flow and bladder emptying.

DETAILED DESCRIPTION:
This study is designed as a multicenter, randomized, controlled, open-label trial. Participants will be randomized 1:1 into two groups using a block randomization method. The experimental group will receive Tamsulosin Hydrochloride Sustained-Release Capsules (0.2 mg, once daily at night) starting 3 days before the biopsy and continuing until the 6th day after the procedure (10 doses total). The control group will not receive Tamsulosin during this perioperative period. All patients will undergo standard pre-biopsy preparations, including bowel preparation and prophylactic antibiotics. The primary endpoint, Acute Urinary Retention (AUR) incidence, along with secondary endpoints (IPSS, QoL, urinary flow rate, post-void residual urine), will be assessed on the 7th day after the biopsy. Safety indicators, such as the incidence of adverse events like orthostatic hypotension and falls, will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 40 to 85 years (inclusive).
* Meets indications for prostate biopsy per clinical guidelines (e.g., suspicious nodule on digital rectal exam, suspicious lesion on imaging, tPSA >10 ng/mL, or tPSA 4-10 ng/mL with f/t <0.16 or PSAD >0.15).
* Voluntarily participates and provides written informed consent.

Exclusion Criteria:

* Previous prostate surgery, urinary diversion, or intermittent catheterization.
* Use of alpha-adrenergic blockers (e.g., Tamsulosin, Doxazosin) within one week prior to screening.
* Known or suspected allergy/intolerance to Tamsulosin, or history of orthostatic hypotension.
* Indwelling urinary catheter or suprapubic cystostomy tube at the time of biopsy.
* History of severe bleeding disorders.
* Poorly controlled or unstable comorbidities such as hypertension or diabetes.
* Severe immunosuppression.
* Severe psychological disorders or uncooperative for the biopsy procedure.
* Active urinary tract infection or neurogenic bladder.
* Any other condition deemed by the investigator as unsuitable for participation.

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1844 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AUR | From biopsy to the 7th day after biopsy.
  Incidence of Acute Urinary Retention (AUR)

SECONDARY OUTCOMES:
IPSS | From baseline (pre-biopsy) to the 7th day after biopsy.
  Change in International Prostate Symptom Score (IPSS)
QoL | From baseline (pre-biopsy) to the 7th day after biopsy.
  Change in Quality of Life (QoL) score related to urinary symptoms
Qmax | From baseline (pre-biopsy) to the 7th day after biopsy.
  Maximum urinary flow rate (Qmax)
PVR | From baseline (pre-biopsy) to the 7th day after biopsy.
  Post-void residual (PVR) urine volume

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Urology Department, Beijing, Outside U.S./Canada, China

IPD SHARING:
Plan to Share IPD: No